CLINICAL TRIAL: NCT01523964
Title: A Phase I, Multi-Center, Controlled, Prospective Correlative Study of Electrical Impedance Myography in Males With Duchenne Muscular Dystrophy and In Healthy Males
Brief Title: DART Electrical Impedance Myography (EIM) Trial in Duchenne Muscular Dystrophy (DMD) and Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dart Therapeutics. LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CMD-001
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; EIM; Duchenne Muscular Dystrophy; electrical impedance myography
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DMD subject ages 3-7 inclusive (Other): Young DMD Testing with EIM
  Interventions: Other: Testing with EIM
- DMD subject ages 8-12 inclusive (Other): Older DMD Testing with EIM
  Interventions: Other: Testing with EIM
- Healthy Control ages 3-7 inclusive (Other): Young Healthy Testing with EIM
  Interventions: Other: Testing with EIM
- Healthy Control ages 8-12 inclusive (Other): Older Healthy Testing with EIM
  Interventions: Other: Testing with EIM

INTERVENTIONS:
Other: Testing with EIM

SUMMARY:
Physicians seek a method to assess neuromuscular disease that is both non-invasive and quantifiable. Many patients do not tolerate standard current day assessment tools (such as needle electromyogram), and Electrical Impedance Myography (EIM) has the potential to serve as a non-invasive, quantifiable, diagnostic tool for neuromuscular disease. If successful, these devices will allow for improved ability to diagnose neuromuscular disease and to assess disease progression or remission, allowing for better care of individual patients as well as for use in clinical trials, where improved outcome measures for neuromuscular diseases is being sought.

DETAILED DESCRIPTION:
Healthy subjects and subjects with DMD will be screened during Visit 1. Screening evaluations will establish eligibility and will include a medical history, abbreviated physical examination, vital signs (blood pressure, temperature, pulse, and respirations), and weight. Eligible subjects will provide assent, as stipulated by Institutional Review Board (IRB) requirements, and a parent/guardian will sign an informed consent, after which the subject will be considered enrolled.

Subjects will be enrolled into 4 study cohorts for a total of approximately 90 subjects. Allocation into these cohorts is planned due to considerations regarding the effect of age on outcomes.

Visit 2, Study Assessments, may take place on the day of Visit 1 screening evaluations. If the subject cannot complete study assessments on the same day, the subject may return and complete Visit 2 evaluations within approximately 24 hours of the end of Visit 1.

Visit 2 assessments will include morphological testing of muscle length and girth, skin fat measurement, Clinical Assessments (6-Minute Walk Test [6MWT], North Star Ambulatory Assessment, timed function tests, dynamometry), and 3 phases of Device Performance testing. Phase 1 Device Performance testing will be done by each of 2 trained raters (Rater A and Rater B) from the research site, designated to perform the Device Performance testing on all subjects at their respective site. At least 10 minutes after completion of the first assessments, Phase 2 Device Performance testing will be repeated by Rater A. Upon completion of the Phase 2 Device Performance testing, the subjects will proceed with Clinical Assessments performed by a physical therapist. Following Clinical Assessments, Phase 3 Device Performance testing will be performed by Rater B.

ELIGIBILITY:
Inclusion Criteria:

DMD Subject Cohorts

* Male subjects
* Subjects with a chronologic age of 3 to 7 years inclusive for Cohort A, and 8 to 12 years inclusive for Cohort B
* Subjects with DMD diagnosed with mutational testing and/or absence of dystrophin on muscle biopsy
* Subjects with proximal pelvic girdle weakness (Gower's maneuver, difficulty with arising from floor and going up steps)
* Subjects who can walk 10 meters unassisted (ie, without braces, canes, or other aids)
* Subjects who are taking systemic corticosteroids and/or any other medication which, in the judgment of the investigator, could impact muscle strength or physical activity levels, must be on a stable dose for at least 4 weeks prior to initiation of study measurements
* Subjects who provide assent, as stipulated by IRB requirements, and whose parent/guardian signs an informed consent form
* Subjects who are willing and able to cooperate and comply with all protocol requirements and procedures

Healthy Control Cohort

* Healthy males with normal neuromuscular examination
* Subjects with a chronologic age of 3 to 7 years inclusive for Cohort C, and 8 to 12 years inclusive for Cohort D
* Subjects who provide assent, as stipulated by IRB requirements, and whose parent/guardian signs an informed consent form
* Subjects who are willing and able to cooperate and comply with all protocol requirements and procedures

Exclusion Criteria:

* Subjects with daytime ventilatory dependence (non-invasive or tracheostomy)
* Subjects enrolled in a DMD therapeutic clinical trial concomitantly or within the past 4 weeks
* Subjects with any physical or mental condition which may, in the investigator's opinion, render the subject unable to complete the tasks of the study appropriately

Ages: 3 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - Massauchusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The University of Texas Southwestern Medical Center-Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from February 2012 to August 2013. Subjects know to the site staff were approached during clinic visits or by telephone to ascertain interest. In addition, referrals from message posted on DMD website were included if they met protocol criteria.
Pre-assignment Details: There were no significant events. Subjects were screened for eligibility and enrolled.
Period: Overall Study
Arm/Group | DMD Subject Ages 3-7 Inclusive | DMD Subject Ages 8-12 Inclusive | Healthy Control Ages 3-7 Inclusive | Healthy Control Ages 8-12 Inclusive
Started | 31 | 30 | 16 | 15
Completed | 31 | 30 | 16 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMD Subject Ages 3-7 Inclusive | DMD Subject Ages 8-12 Inclusive | Healthy Control Ages 3-7 Inclusive | Healthy Control Ages 8-12 Inclusive | Total
Number analyzed (Participants) | 31 | 30 | 16 | 15 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 30 | 16 | 15 | 92
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 31 | 30 | 16 | 15 | 92
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 16 | 15 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Adverse Event.
Description: Adverse events will be assessed during the time the subject is enrolled in the trial.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | DMD Subject Ages 3-7 Inclusive | DMD Subject Ages 8-12 Inclusive | Healthy Control Ages 3-7 Inclusive | Healthy Control Ages 8-12 Inclusive
Number analyzed (Participants) | 31 | 30 | 16 | 15
participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day (length of subject participation)
Arm/Group | DMD Subject Ages 3-7 Inclusive | DMD Subject Ages 8-12 Inclusive | Healthy Control Ages 3-7 Inclusive | Healthy Control Ages 8-12 Inclusive
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/31 | 0/30 | 0/16 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DMD Subject Ages 3-7 Inclusive (N=31) | DMD Subject Ages 8-12 Inclusive (N=30) | Healthy Control Ages 3-7 Inclusive (N=16) | Healthy Control Ages 8-12 Inclusive (N=15)
scab on left ankle abrasion dislodged (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Subject has prior left ankle abrasion with scab. During 6 minute walk scab was dislodged during a fall.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less